CLINICAL TRIAL: NCT05678335
Title: Tacrolimus for Mild Thrombocytopenia in Sjogren's Syndrome
Brief Title: Tacrolimus for Thrombocytopenia in SS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Prof., Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-22PJ1065
Record Dates: First submitted 2022-12-28; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Sjogren Syndrome With Other Organ Involvement
Keywords: Sjogren's syndrome; Thrombocytopenia; Tacrolimus
MeSH Terms: conditions — Sjogren's Syndrome; Thrombocytopenia | interventions — Hydroxychloroquine; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine monotherapy (Placebo Comparator): Oral hydroxychloroquine 200mg twice daily for 12 weeks.
  Interventions: Drug: Hydroxychloroquine
- Tacrolimus monotherapy (Experimental): Oral tacrolimus 1-2mg twice daily for 12 weeks.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Hydroxychloroquine — Oral hydroxychloroquine 200mg twice daily for 12weeks.
  Arms: Hydroxychloroquine monotherapy
Drug: Tacrolimus — Oral Tacrolimus 1-2mg twice daily for 12 weeks.
  Arms: Tacrolimus monotherapy

SUMMARY:
This 12-week randomized, open-label study evaluates the efficacy and safety of Tacrolimus for Sjogren's syndrome patients with thrombocytopenia.

DETAILED DESCRIPTION:
This study evaluates the efficacy and safety of Tacrolimus for the treatment of thrombocytopenia in Sjogren's syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Sjogren's syndrome according to the 2002 revised American-European Consensus Group (AECG) criteria.
* Baseline platelet counts within 30-80×109/L.

Exclusion Criteria:

* Concomitant other systemic autoimmune diseases.
* Severe complications of Sjogren's syndrome.
* Abnormal laboratory tests such as: white blood cell count <2.5x10^9/L, hemoglobin <80 g/L, AST/ALT >1.5 ULN, serum creatine > 1.5 mg/dL.
* Received glucocorticoids, immunosuppressants, or biological agents within 3 months.
* Active acute or chronic infections.
* History of malignancy.
* Pregnancy or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | week 12
  Complete response (platelet counts > 100×10^9/L) rates at week 12.

SECONDARY OUTCOMES:
Complete response rate | week 4 and week 8
  Complete response (platelet counts > 100×10^9/L) rates at week 4 and week 8.
ESSDAI improvement | week 12
  Change from baseline in ESSDAI (EULAR Sjogren's Syndrome Disease Activity Index) score at week 12.
ESSPRI improvement | week 12
  Change from baseline in ESSPRI (EULAR Sjogren's Syndrome Patient Reported Index) score at week 12.

OTHER OUTCOMES:
Immunoglobulins | week 12
  Change from baseline in Immunoglobulin (IgG, IgM and IgA) levels at week 12.
Rheumatoid Factor | week 12
  Change from baseline in rheumatoid factor level at week 12.

IPD SHARING:
Plan to Share IPD: Undecided